CLINICAL TRIAL: NCT03553615
Title: Open-label Pilot Clinical Trial of Oral Ivermectin to Treat Atopic Dermatitis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Limited clinical capacity
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Kavita Sarin, Assistant Professor of Dermatology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-46486
Record Dates: First submitted 2018-05-30; First posted 2018-06-12 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Ivermectin

STUDY DESIGN:
Intervention Model Description: Oral Ivermectin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Oral treatment (Experimental): 12mg oral ivermectin treatment taken once a week for four weeks
  Interventions: Drug: Ivermectin Pill

INTERVENTIONS:
Drug: Ivermectin Pill — oral anti-parasitic agent taken as a weekly dose for four weeks
  Other Names: Stromectol

SUMMARY:
This pilot trial studies how well a novel oral therapeutic agent performs to treat patients with atopic dermatitis, particularly facial dermatitis.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Overall response rate of atopic dermatitis in subjects as assessed using Dermatology Life Quality Index (a 10 question questionnaire used to measure the impact of skin disease on the quality of life of an affected person)

SECONDARY OBJECTIVES:

I. , Eczema Area and Severity Index (EASI), Total Severity Scoring (TSS) II. Safety assessment after 8 weeks with 4 weeks of oral treatment. III. VAS (Visual Analogue Scale, an instrument for the assessment of pruritus) at baseline through eight weeks.

OUTLINE:

Patients receiving novel oral agent once a week for 4 weeks in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Must have at least one lesion of atopic dermatitis (At least 1% Body surface Area).
2. 18 years of age or older.
3. Must be willing to take oral ivermectin once weekly for 4 weeks and monitor over 8 weeks.
4. For women of child bearing potential, a negative urine pregnancy test
5. Women of child bearing potential are expected to use an effective method of birth control while participating in the study and for 1 month after taking the last dose.
6. For male subjects with female partners of childbearing potential, agreement to use adequate contraception while participating in the study and for 1 month after taking the last dose.
7. Has signed and dated the current Institutional Review Board approved informed consent document.
8. Must be able to read and speak English fluently.

Exclusion Criteria:

1. Is currently participating or has participated in another interventional clinical study in the past 2 weeks;
2. Is age <18 years old.
3. Has had known or previous hypersensitivity or allergic reactions to oral ivermectin before;
4. Has an immunologic or infectious disease (e.g. hepatitis, tuberculosis, HIV or AIDS, lupus rheumatoid arthritis) which could place the subject at risk or interfere with the accuracy of the study results;
5. Taking any medication known to interact with ivermectin like Dasabuvir (theoretical) or warfarin (probable).
6. Is planning a trip to a sunny climate, to use tanning booths or use other UV sources throughout the course of this study;
7. Has a history of hypersensitivity to any substance in investigational preparation;
8. Has any clinically significant medical condition or laboratory abnormality that would, in the opinion of the Investigator, put the patient at undue risk or interfere with the interpretation of the study results;
9. Is currently pregnant or breastfeeding.
10. Has other skin conditions that might interfere with Atopic Dermatitis diagnosis and/or evaluation (i.e. psoriasis current active viral, bacterial and fungal skin infections) as assessed by the Investigator;
11. Any other condition or factor the Investigator or their duly assigned representative believes may affect the ability of the subject to complete the study or the interpretation
12. History of congestive heart failure; cardiac arrhythmias; or other findings of ventricular dysfunction.
13. History of current evidence of malabsorption or liver disease.
14. Cannot read and speak English fluently.
15. Does not have at least 1% body surface area with lesional atopic dermatitis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2030-12-01 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
DLQI | 8 weeks
  Patient Dermatology Life Quality Index

SECONDARY OUTCOMES:
EASI | 8 weeks
  Eczema area and severity index
TSS | 8 weeks
  Total Sum Score of lesion
IGA | 8 weeks
  Investigator Global Analysis
VAS for Pruritis | 8 weeks
  Visual Analogue Scale for Pruritis

CONTACTS AND LOCATIONS:
Overall Officials: Kavita Sarin, MD, PhD, Study Director — Stanford University
Locations (1):
- Stanford Hospital and Clinics, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No